CLINICAL TRIAL: NCT05474495
Title: Comparative Effects of Transversus Abdominis and Pelvic Floor Muscle Strengthening Exercise Program on Disability and Urinary Incontinence In Patients With Grade 1 Cystocele
Brief Title: Transversus Abdominis and Pelvic Floor Muscle Strengthening Exercise Program In Patients With Grade 1 Cystocele
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0533
Record Dates: First submitted 2022-07-24; First posted 2022-07-26 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Disability Physical; Urinary Incontinence; Prolapse
Keywords: Cystocele; Disability; Pelvic Floor Prolapse; Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence; Prolapse; Cystocele

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pelvic floor muscle training (Experimental): Experimental Group (Group A) will receive pelvic floor muscle training. Two sessions a week for 6 weeks, each session lasting 45 mins.
  Interventions: Other: Pelvic floor muscle training
- Transverse abdominas strength training (Active Comparator): Active Comparator (Group B) will receive transverse abdominas strength training. Treatment will be given 5 days a week and continued for 6 weeks.
  Interventions: Other: Transverse abdominas strength training

INTERVENTIONS:
Other: Pelvic floor muscle training — Pelvic floor muscle training. Two sessions a week for 6 weeks, each session lasting 45 mins.
  Arms: Pelvic floor muscle training
Other: Transverse abdominas strength training — Transverse abdominas strength training will be given 5 days a week and continued for 6 weeks.
  Arms: Transverse abdominas strength training

SUMMARY:
Cystocele, a protrusion of the bladder, happens while the bladder descends into the vagina. There are more than one underlying causes for the development of cystocele ensuing in weak point of the muscles and the connective tissue surrounding the bladder and vagina.

This study will be a randomized clinical trial. After the department permission of physical therapy data will be collected from patient of Jinnah Hospital. Data will be collected before and after treatment. Randomization will be done by lottery method. Group A will be given pelvic floor strengthning exercises and goup B will be given transverse abdominas strengthning exercises. Each group will have 33 patients each. A 6-week physical therapy program will be planned. Group A will be given pelvic floor muscle strengthning exercise and the group B will given transverse abdominas exercises.Data will be entered and analysed by SPSS version 25.

DETAILED DESCRIPTION:
Cystocele, in any other case called a protrusion of the bladder, happens while the bladder descends into the vagina.The bladder bulges via the anterior wall of the vagina, with which it's miles anatomically related. There are more than one underlying causes for the development of cystocele ensuing in weak point of the muscles and the connective tissue surrounding the bladder and vagina. This study will be a randomized clinical trial. After the department permission of physical therapy data will be collected from patient of Jinnah Hospital. Data will be collected before and after treatment. Total sample size is 60. Non probability convenient sampling technique will be used. Randomization will be done by lottery method. Group A will be given pelvic floor strengthning exercises and goup B will be given transverse abdominas strengthning exercises. Each group will have 33 patients each. A 6-week physical therapy program will be planned. Group A will be given pelvic floor muscle strengthning exercise and the group B will given transverse abdominas exercises. Individual sessions will be held twice a week for 60 minutes each. Each meeting will include a theoretical portion of up to 10 minutes and a practical portion of roughly 50 minutes. Home plan will also be shared with them. Post treatment analysis will be done in order to find the effects of both regims. Data will be entered and analysed by SPSS version 25. The aim is to compare the effects of transversus abdominis and pelvic floor muscle strengthening exercise program on disability and urinary incontinence in patients with grade 1 cystocele.

ELIGIBILITY:
Inclusion Criteria:

* Females age of 35 to 65 years will be included in our study.
* Females who will not able to contract the Pelvic floor muscles
* Female who hill have mixed urinary incontinence will be included in our study

Exclusion Criteria:

* Females with malignancies will be excluded
* Females with neurological issue will be excluded
* Females who hill have untreated urinary tract infection will be excluded from our study

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females With Grade 1 Cystocele
Enrollment: 60 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Pelvic Floor Disability Index | 6 Weeks
  The Pelvic Floor Disability index Questionnaire is a condensed version of the Pelvic Floor Distress Inventory (PFDI).The PFDI-20 has 20 items and 3 scales of your symptoms. All items use the following format with a response scale from 0 to 4. Scale Scores: Obtain the mean value of all of the answered items within the corresponding scale (possible value 0 to 4) and then multiply by 25 to obtain the scale score (range 0 to 100).
Pelvic organ prolapse quantification (POP-Q) | 6 Weeks
  It will be used for diagnostic purpose for prolapse and participants will only be considered as Grade 1 Cystocele on the basis of this tool. and it will also used to compare the Exercise effects on prolapse at the start and at the end of study. It uses objective and precise distance measurements to the reference point, the hymen. Cystocele and prolapse of the vagina from other causes is staged using POP-Q criteria and can range from good support (no descent into the vagina) reported as a POP-Q stage 0 or I to a POP-Q score of IV, which includes prolapse beyond the hymen. It also used to quantify the movement of other structures into the vaginal lumen and their descent.

CONTACTS AND LOCATIONS:
Overall Officials: Sabiha Arshad, M.Phil, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital,, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muro S, Tsukada Y, Harada M, Ito M, Akita K. Anatomy of the smooth muscle structure in the female anorectal anterior wall: convergence and anterior extension of the internal anal sphincter and longitudinal muscle. Colorectal Dis. 2019 Apr;21(4):472-480. doi: 10.1111/codi.14549. Epub 2019 Jan 24. PMID 30614646
- [Background] Roch M, Gaudreault N, Cyr MP, Venne G, Bureau NJ, Morin M. The Female Pelvic Floor Fascia Anatomy: A Systematic Search and Review. Life (Basel). 2021 Aug 30;11(9):900. doi: 10.3390/life11090900. PMID 34575049
- [Background] Flusberg M, Kobi M, Bahrami S, Glanc P, Palmer S, Chernyak V, Kanmaniraja D, El Sayed RF. Multimodality imaging of pelvic floor anatomy. Abdom Radiol (NY). 2021 Apr;46(4):1302-1311. doi: 10.1007/s00261-019-02235-5. PMID 31555847
- [Background] Stupart D, Pickles K, Briggs C. Anatomy of the vesicovaginal fascia and its relation to branches of the inferior hypogastric plexus. Clin Anat. 2022 Oct;35(7):855-860. doi: 10.1002/ca.23858. Epub 2022 Apr 2. PMID 35333406
- [Background] Eid S, Iwanaga J, Oskouian RJ, Loukas M, Tubbs RS. Comprehensive Review of the Cardinal Ligament. Cureus. 2018 Jun 20;10(6):e2846. doi: 10.7759/cureus.2846. PMID 30140597